CLINICAL TRIAL: NCT04657289
Title: A Phase IIIb, Global, Multicenter, Randomized, Visual Assessor-Masked Study of the Efficacy, Safety, and Pharmacokinetics of a 36-Week Refill Regimen for the Port Delivery System With Ranibizumab in Patients With Neovascular Age-Related Macular Degeneration (Velodrome)
Brief Title: A Study of the Efficacy, Safety, and Pharmacokinetics of a 36-Week Refill Regimen for the Port Delivery System With Ranibizumab in Patients With Neovascular Age-Related Macular Degeneration (Velodrome)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WR42221; 2020-001313-20 (EudraCT Number); CIV-21-02-035827 (Other: EUDAMED NUMBER); 2023-507130-24-00 (EU CTIS Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD)
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Intervention Model Description: Phase 3b
Who Masked: Outcomes Assessor
Masking Description: * The BCVA examiner will only conduct refraction and BCVA assessments and will be masked to participant study eye assignment and study visit type.
  * The BCVA examiner will have no access to a participant's BCVA scores from previous visits and will be aware only of the participant's refraction data from previous visits.
  * The BCVA examiner may provide no other direct or indirect participant care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Arm A [Q36W] 36-weeks between refill-exchange procedures (Experimental): Participants randomized to the Q36W arm will receive PDS implant refill-exchange procedures (ranibizumab 100 mg/mL) on a Q36W fixed interval.
  Interventions: Drug: Ranibizumab; Device: Port Delivery System with Ranibizumab
- Arm B [Q24W] 24-weeks between refill-exchange procedures (Active Comparator): Participants randomized to the Q24W arm will receive PDS implant refill-exchange procedures (ranibizumab 100 mg/mL) on a Q24W fixed interval.
  Interventions: Drug: Ranibizumab; Device: Port Delivery System with Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Arm A: Participants will receive ranibizumab delivered through the PDS implant with 100 mg/mL in the study eye on Day 1 and receive refill-exchanges at fixed 36-week intervals
  Arm B: Participants will receive ranibizumab delivered through the PDS implant with 100 mg/mL in the study eye on Day 1 and receive refill-exchanges at fixed 24-week intervals
Device: Port Delivery System with Ranibizumab — Arm A: Participants will receive ranibizumab delivered through the PDS implant with 100 mg/mL in the study eye on Day 1 and receive refill-exchanges at fixed 36-week intervals
  Arm B: Participants will receive ranibizumab delivered through the PDS implant with 100 mg/mL in the study eye on Day 1 and receive refill-exchanges at fixed 24-week intervals

SUMMARY:
Study WR42221 is a Phase IIIb, global, multicenter, randomized, visual assessor-masked study designed to assess the efficacy, safety, and pharmacokinetics of the Port Delivery System with ranibizumab (PDS) 100 mg/mL delivered every 36 weeks (Q36W) compared with every 24 weeks (Q24W) in patients with neovascular age-related macular degeneration (nAMD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years at time of signing Informed Consent Form
* Initial diagnosis of nAMD within 9 months prior to the screening visit
* Previous treatment with at least three anti- vascular endothelial growth factor (VEGF) intravitreal injections for nAMD per standard of care within 6 months prior to the screening visit
* Demonstrated response to prior anti-VEGF intravitreal treatment since diagnosis
* Availability of historical visual acuity data prior to the first anti-VEGF treatment for nAMD until the time of study enrollment
* BCVA of 34 letters (approximate 20/200 Snellen equivalent) or better

Exclusion Criteria:

* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in study eye
* Prior treatment with Visudyne®, external-beam radiation therapy, or transpupillary thermotherapy in study eye
* Previous treatment with corticosteroid intravitreal injection, intraocular device implantation, previous laser (any type) used for AMD treatment in study eye
* Treatment with anti-VEGF agents other than ranibizumab within 1 month prior to the enrollment visit in study eye
* Concurrent conjunctival, Tenon's capsule, and/or scleral condition in the supero-temporal quadrant of the eye that may affect the implantation, subsequent tissue coverage, and refill-exchange procedure of the PDS implant
* Prior treatment with brolucizumab (at any time prior to the screening visit) in either eye
* Prior participation in a clinical trial involving any anti-VEGF drugs, within 9 months prior to the enrollment visit in either eye
* Subretinal hemorrhage that involves the center of the fovea, if the hemorrhage is >0.5 disc area at screening in study eye
* Subfoveal fibrosis or subfoveal atrophy in study eye
* Choroidal neovascularization (CNV) due to other causes, such as ocular histoplasmosis, trauma, central serous chorio-retinopathy, or pathologic myopia in either eye
* Retinal pigment epithelial tear in study eye
* Any concurrent intraocular condition that would either require surgical intervention during the study to prevent or treat visual loss that might result from that condition or affect interpretation of study results in study eye
* Active intraocular inflammation in study eye
* History of vitreous hemorrhage in study eye
* History of rhegmatogenous retinal detachment in study eye
* History of retinal tears or peripheral retinal breaks within 3 months prior to the enrollment visit in study eye
* History of pars plana vitrectomy surgery
* Aphakia or absence of the posterior capsule in study eye
* Spherical equivalent of the refractive error demonstrating more than 8 diopters of myopia in study eye
* Preoperative refractive error that exceeded 8 diopters of myopia, for Participants who have undergone prior refractive or cataract surgery in study eye
* Intraocular surgery within 3 months preceding the enrollment visit in study eye
* Uncontrolled ocular hypertension or glaucoma and any such condition the investigator determines may require a glaucoma-filtering surgery during a participant's participation in the study in study eye
* History of glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery in study eye
* History of corneal transplant in study eye
* Any history of uveitis requiring treatment in either eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled blood pressure
* History of stroke within the last 3 months prior to informed consent
* Atrial fibrillation diagnosed or worsened within the last 3 months prior to informed consent
* History of myocardial infarction within the last 3 months prior to informed consent,
* History of other disease, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of ranibizumab or placement of the implant and that might affect interpretation of the results of the study or renders the participant at high risk of treatment complications in the opinion of the investigator
* Confirmed active systemic infection
* Use of any systemic anti-VEGF agents
* Active cancer within 12 months of enrollment except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, and prostate cancer with a Gleason score of <= 6 and a stable prostate-specific antigen for > 12 months
* Previous participation in any non-ocular disease studies of investigational drugs within 1 month preceding the informed consent
* Non-functioning non-study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2027-01-07 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Best-corrected visual acuity (BCVA) score averaged over Weeks 68 and 72, as assessed using the ETDRS chart starting at a distance of 4 meters | Baseline to Week 72
  EDTRS = Early Treatment Diabetic Retinopathy Study. A vision score of 20/20 vision is considered normal. A score of 20/200 is considered being legally blind.

SECONDARY OUTCOMES:
Change from baseline in BCVA score over time | Baseline up to Week 72
Percentage of participants with BCVA score of 69 letters (approximate 20/40 Snellen equivalent) or better averaged over Weeks 68 and 72 | Baseline to Week 72
Percentage of participants with BCVA score of 69 letters (approximate 20/40 Snellen equivalent) or better over time | Baseline up to Week 72
Percentage of participants with BCVA score of 38 letters (approximate 20/200 Snellen equivalent) or worse averaged over Weeks 68 and 72 | Baseline to Week 72
Percentage of participants with BCVA score of 38 letters (approximate 20/200 Snellen equivalent) or worse over time | Baseline up to Week 72
Percentage of participants who report preferring ranibizumab 100 mg/mL delivered via the PDS compared with intravitreal treatment, as measured by the PDS Patient Preference Questionnaire (PPPQ) at At Weeks 24, 40 and 72 | At Weeks 24, 40, 72
Percentage of participants with bilateral disease who report preferring ranibizumab 100 mg/mL delivered via the PDS compared with intravitreal treatment, as measured by the PPPQ at At Weeks 24, 40 and 72 | At Weeks 24, 40, 72
Mean overall treatment satisfaction at Week 40, as measured by the Macular Disease Treatment Satisfaction Questionnaire (MacTSQ) total score in the Q36W arm compared with the Q24W arm | At Week 40
Percentage of participants who lose <10, <5, or gain >= 0 letters in BCVA score from baseline averaged over Weeks 68 and 72 | Baseline to Week 72
Percentage of participants who lose <10, <5, or gain >= 0 letters in BCVA score from baseline over time | Baseline up to Week 72
Incidence and severity of ocular and systemic (non-ocular) adverse events in the Q36W and Q24W arms | Baseline up to Week 72
Incidence, severity, and duration of adverse events of special interest, including ocular adverse events of special interest in the Q36W and Q24W arms | Baseline up to Week 72
Incidence, severity, and duration of ocular adverse events of special interest during the postoperative period (≤ 37 days of initial implantation) and follow-up period (> 37 days after implantation surgery) in all enrolled participants | Baseline up to Week 72
Incidence and severity of adverse device effects in the Q36W and Q24W arms | Baseline up to Week 72
Incidence, causality, severity, and duration of anticipated serious adverse device effects in the Q36W and Q24W arms | Baseline up to Week 72
Change from baseline in center point thickness (CPT) up to and including Week 72 | Baseline up to Week 72
Percentage of participants who do not undergo supplemental treatment with intravitreal ranibizumab 0.5 mg before each refill-exchange procedure | Week 16 to Week 68
Observed serum concentration of ranibizumab at specified timepoints | Baseline to Week 72
Incidence of treatment-emergent ADAs during the study | Baseline to Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (108):
- Argentina (3):
  - Centro Oftalmologico Dr. Charles S.A., Capital Federal
  - Oftalmos, Capital Federal
  - Grupo Laser Vision, Rosario
- Australia (10):
  - Eyeclinic Albury Wodonga, Albury, New South Wales
  - Eye and Retina Consultants, Hurstville, New South Wales
  - Retina Associates Liverpool, Liverpool, New South Wales
  - Retina and Macula Specialists, Miranda, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Queensland Eye Institute, Woolloongabba, Queensland
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- Austria (2):
  - LKH-Univ.Klinikum Graz, Graz
  - Medizinische Universitat Wien, Vienna
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Brazil (6):
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Botelho Hospital da Visao, Blumenau, Santa Catarina
  - Retina Clinic, São Paulo, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESPX, São Paulo, São Paulo
  - Instituto da Visao IPEPO, São Paulo, São Paulo
  - Hosp de Olhos de Sorocaba, Sorocaba, São Paulo
- France (7):
  - Centre Retine Gallien, Bordeaux
  - Hopital de la croix rousse, Lyon
  - Centre Paradis Monticelli, Marseille
  - CHU Nantes - Hotel Dieu, Nantes
  - Hopital Lariboisiere, Paris
  - Fondation Rothschild, Paris
  - Hopital PURPAN - CHU TOULOUSE, Toulouse
- Germany (12):
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinikum Koln, Cologne
  - Medizinische Universitat Lausitz ? Carl Thiem, Cottbus
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - LMU Klinikum der Universitat, Augenklinik, München
  - Augenabteilung am St. Franziskus-Hospital, Münster
  - Universitatsklinikum Munster, Münster
  - Knappschaftsklinikum Saar GmbH, Sulzbach
  - Universitatsklinikum Tubingen, Tübingen
  - Universitatsklinikum Ulm, Augenklinik und Poliklinik, Ulm
- Israel (6):
  - Rambam Medical Center, Haifa
  - Hadassah MC, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin MC, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky MC, Tel Aviv
- Italy (13):
  - Ospedale Clinicizzato SS Annunziata, Chieti, Abruzzo
  - Policlinico di Bari, Bari, Apulia
  - Azienda Ospedaliero Universitaria "Ospedali Riuniti" Trieste-Ospedale Maggiore, Trieste, Friuli Venezia Giulia
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Fondazione G.B. Bietti Per Lo Studio E La Ricerca in Oftalmologia-Presidio Ospedaliero Britannico, Rome, Lazio
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico-Clinica Regina Elena, Milan, Lombardy
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Asst Fatebenefratelli Sacco, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette - Ancona, The Marches
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera di Perugia Ospedale S. Maria Della Misericordia, Perugia, Umbria
  - Ospedale Classificato Equiparato Sacro Cuore ? Don Calabria, Negrar - Verona, Veneto
  - A.O. Universitaria S. Maria Della Misericordia Di Udine, Udine, Veneto
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore Eye Research Institute, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (9):
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Kim's Eye Hospital, Seoul
- Spain (12):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, San Cugat Del Valles, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Instituto Oftalmologico Fernandez Vega, Oviedo, Principality of Asturias
  - Centro de Oftalmologia Barraquer, Barcelona
  - Institut de la Macula i la retina, Barcelona
  - Hospital dos de maig, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Arruzafa. Servicio de Oftalmologia, Córdoba
  - Clinica Baviera, Madrid
  - Oftalvist Valencia, Valencia
- Switzerland (5):
  - Universitatsspital Basel Augenklinik Klinik, Basel
  - Inselspital Bern Ophthalmologische Klinik, Bern
  - Vista Klinik Ophthalmologische Klinik, Binningen
  - Fondation Asile Des Aveugles ? Jules Gonin Eye Hospital, Lausanne
  - Stadtspital Triemli Ophthalmologische Klinik, Zurich
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
  - National Taiwan University Hospital, Zhongzheng Dist.
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Ankara Etlik City Hospital, Ankara
  - Beyoglu Goz Training and Research Hospital, Istanbul
  - Kocaeli Universitesi T?p Fakultesi, Kocaeli
- United Kingdom (9):
  - Bristol Eye Hospital, Bristol
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Central Middlesex Hospital, London
  - Kings College Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Sunderland Eye Infirmary, Sunderland
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing